CLINICAL TRIAL: NCT03273998
Title: Cross-sectional Study on Prevalence of Coagulation Factors Deficiency in Children Attending Assiut University Children Hospital ( a One Year Study)
Brief Title: Cross-sectional Study on Prevalence of Coagulation Factors Deficiency in Assiut University Children Hospital
Acronym: coagdef
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, YHAlattar, principle investigator, Assiut University
Other Study IDs: Coag Def
Record Dates: First submitted 2017-08-29; First posted 2017-09-06 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Coagulation Factor Deficiency
Keywords: coagulation; bleeding
MeSH Terms: conditions — Thrombosis; Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Blood coagulation is a complex mechanism that is required for the rapid establishment of a stable fibrin clot. A series of interdependent enzyme-mediated reactions translate the molecular signals that initiate blood coagulation into the formation of the fibrin clot. Congenital coagulopathies result when there is a deficiency of protein co factors and enzymes implicated in blood coagulation

DETAILED DESCRIPTION:
The most frequent inherited coagulation disorders are haemophilia A and B, due to the deﬁciency of factor VIII and IX. Haemophilia A and B are clinically indistinguishable from each other and occur in mild, moderate and severe forms (with plasma factor levels of 6-30%, 2-5% and 1% or less respectively). Inherited as X-linked traits, haemophilia A and B are prevalent in the general population of approximately 1 in 10 000 and 1 in 50 000, with no signiﬁcant racial difference. Other deﬁciencies of coagulation factors that cause a bleeding disorder, such as aﬁbrinogenaemia, hypoprothrombinaemia, deﬁciencies of factors V and combined factor V and VIII, VII, X, XI and XIII are inherited as autosomal recessive traits and are generally much rarer than the haemophilias, wich are prevalent in the general population varying between 1 in 500 000 and 1 in 2 000 000. As a consequence of the rarity of these deﬁciencies, which are expressed clinically only in homozygotes or compound heterozygotes, the type and severity of symptoms, the underlying molecular defects and the actual management of bleeding episodes are not well established as for haemophilia A and B.

Inherited deficiencies are described for all of the known coagulation factors. In addition, there are people with an abnormal bleeding tendency for whom no cause has yet been identified. The concept of overall hemostatic balance is increasingly recognized, that it is not solely the level of a single factor that matters, but the overall control of hemostasis that may determine the bleeding risk. This may explain why the bleeding risk cannot be predicted from a single factor level alone as in, for example, factor VII or factor XI deficiency in particular. The rare factor deficiencies have several common properties: they are inherited in an autosomal manner, although bleeding symptoms have been described in heterozygous partially deficient individuals. These rare deficiencies are more common in populations and countries where cousin marriages are frequent and therefore there is considerable geographic variation in the incidence, in contrast to hemophilia and von Willebrand disease types I or II which occur with the same incidence in different countries.

Clinical manifestations:

In their most severe form, the deficiencies present with serious hemorrhage in the neonatal period; intracranial hemorrhage is a significant presentation of severe deficiency of FXIII, factor VII, factor X or fibrinogen (afibrinogenaemia). Bleeding from the umbilical stump can occur with any of these disorders as it can with severe hemophilia. It is important for caregivers to be aware that any unusual bleeding manifestation must prompt appropriate investigation so that diagnosis is not delayed, and appropriate replacement therapy is given as soon as possible. A history of consanguinity of the parents and their ethnic origin are relevant.

Diagnosis should be straightforward but there are pitfalls in testing. Difficult venepunctures in infants in an emergency may give erroneous results due to tissue factor contamination. Coagulation samples do not travel well, so if plasma samples are sent to another laboratory they must be properly transported, generally frozen and sent on dry ice. It may be helpful to test both parents because, apart from the two truly recessive disorders detailed below, the parents will usually have evidence of partial deficiency. It is important for each laboratory to establish its own normal range, and to ensure that the possibility of genetic carriage of a disorder is fully discussed with parents irrespective of the blood results as the birth of more children with a serious bleeding disorder is a great emotional and social burden especially in countries and communities with poor health resources.

Fibrinogen deficiency

Fibrinogen deficiency is heterogeneous and two main phenotypes can be distinguished. In afibrinogenaemia, plasma and platelet levels of the protein are unmeasurable or very low when using assays that measure clottable and immunoreactive protein, whereas in dysfibrinogenaemia low clottable fibrinogen contrasts with normal or moderately reduced fibrinogen antigen.

Clinical manifestations:

Whereas most patients with dysfibrinogenaemia do not bleed at all, afibrinogenaemic patients have a bleeding tendency.

Among severe bleeding symptoms that are dangerous for life and for the musculoskeletal function, umbilical cord and joint bleeding is relatively frequent (in 75% and 50% of patients), whereas muscle hematomas and bleeding in the gastrointestinal tract and central nervous system are less common.

Milder symptoms such as epistaxis and menorrhagia are also frequent. Post-partum bleeding occurs when no prophylactic replacement therapy is given. Excessive blood loss and impaired wound healing in about one-third of the patients often accompany circumcision and other surgical maneuvers. There is no increased prevalence of recurrent miscarriages. Central nervous system bleeding is rare.

Factor V deficiency Congenital factor V deficiency (also known as labile factor or proaccelerin) is a rather uncommon [1:1000,000] inherited coagulopathy (autosomal recessive inheritance).

Affected patients become symptomatic in early childhood with spontaneous or post- traumatic bleeding complications

Factor VII deficiency

Factor VII deficiency is the most common autosomal recessive coagulation disorder (1 per 500 000 population). Factor VII circulates in plasma at a concentration of approximately 0.5 μg/mL (10 mmol/L). Plasma levels of factor VII coagulant activity (FVII:C) and FVII antigen (FVII: Ag) are influenced by a number of genetic and environmental factors (sex, age, cholesterol and triglyceride levels). The majority of patients have concomitantly low levels of factor VII functional activity and antigen, but several cases are characterized by normal or low borderline levels of factor VII antigen, contrasting with lower levels of functional activity. Most gene knockout mice made experimentally deficient in factor VII develop normally but some suffer fatal perinatal bleeding.

Clinical manifestations:

The severity of symptoms of factor VII deficiency is variable and generally reported to be poorly correlated with plasma levels. Some patients do not bleed at all after major challenges of haemostasis, and even cases of thrombosis have been described. life- or limb-endangering bleeding manifestations are relatively rare, the most frequent symptoms being epistaxis and menorrhagia. However, the prevalence of haemarthroses and soft-tissue bleeding was less than that found in other large series. The risk of central nervous system bleeding in infants with severe factor VII deficiency is high in some series.

Factor VIII & factor IX deficiency:

The hemophilias are X-linked congenital bleeding disorders, and the two major categories are hemophilia A (factor VIII deficiency, seen in 1 in 5,000 male births) and hemophilia B (factor IX deficiency, seen 1 in 30,000 male births) Prophylaxis for children with severe hemophilia consists of infusion of a factor concentrate two or three times a week in order to keep blood levels of factor VIII or IX high enough to prevent bleeding. On-demand therapy involves infusion of a factor concentrate immediately after bleeding starts in an effort to prevent joint or muscle damage

Factor XI deficiency Factor XI deficiency is characterized by a decrease of the functional activity of this plasma protein, usually accompanied by correspondingly low levels of factor XI antigen. Most of cases reported in the literature are of Ashkenazi Jewish origin, the frequency of heterozygosity for factor XI deficiency being as high as 8% in this population. In knockout mice, the loss of the gene coding for this factor is compatible with life, with no tendency for spontaneous bleeding.

Clinical manifestations:

The relationship between the residual factor XI levels in plasma and the bleeding tendency is not as clear-cut as for other coagulation factor deficiencies. Usually, patients with severe factor XI deficiency (1% or less) are mildly affected and have bleeding symptoms only after trauma or surgery. Surprisingly patients with low but detectable levels of factor XI are also mild bleeders, severe or moderate deficiency (factor XI < 1-5%) and in patients with mild deficiency (6-30%). All patients were mild bleeders, but those symptoms that define the severity of the bleeding tendency, such as muscle hematomas and hemarthroses, showed a similar frequency in the two groups of deficient patients (approximately 25%). The most frequent symptoms were oral and post-operative bleeding, which occurred in more than 50% of patients.

Differential diagnosis :

Causes of congenital bleeding disorders

The most common include:

Von Willebrand Disease Hemophilia A (Factor Viii Deficiency) Hemophilia B(Factor Ix Deficiency)

Less Common :

Factor 1(Fibrinogen Deficiency) Factor II (Prothrombin Deficiency or Dysfunction) Factor V Deficiency Factor VII Deficiency Factor X Deficiency Factor XI Deficiency Factor XIII Deficiency Platelet Disorders Congenital Aplastic Anemia

ELIGIBILITY:
Inclusion Criteria:

* All patients with congenital bleeding disorders secondary to coagulation factor deficiency and attending in Assiut University Children Hospital will be included in the study

Exclusion Criteria:

* Patients with:

Acquired bleeding disorders Thrombasthenia thrombocytopenia

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children with coagulation factors deficiency in Assiut University Children Hospital
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
prevalence of children with coagulation factors deficiency in Assiut University Children Hospital measured by coagulation factor deficiency checklist | 1year
  data collected in sheet measuring type and level of deficient factor and measuring clotting tests(e.g. pt ,aptt)

SECONDARY OUTCOMES:
evaluation of inheritance of coagulation fa tors deficiency through the checklist measuring other affected family members | 1year
  number of family members having coag factors deficiency , their age ,sex
evaluation of infectious disease by measuring hepatitis c virus and human immunodeficiency virus | one year
  hepatitis c virus and human immunodeficiency virus testing

CONTACTS AND LOCATIONS:
Overall Officials: yomna alattar, resident, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mannucci PM, Duga S, Peyvandi F. Recessively inherited coagulation disorders. Blood. 2004 Sep 1;104(5):1243-52. doi: 10.1182/blood-2004-02-0595. Epub 2004 May 11. PMID 15138162
- [Result] Bolton-Maggs PH. The rare inherited coagulation disorders. Pediatr Blood Cancer. 2013;60 Suppl 1:S37-40. doi: 10.1002/pbc.24336. Epub 2012 Oct 25. PMID 23109366
- [Result] Peyvandi F, Mannucci PM. Rare coagulation disorders. Thromb Haemost. 1999 Oct;82(4):1207-14. PMID 10544899
- [Result] Ehrenforth S, Klarmann D, Zabel B, Scharrer I, Kreuz W. Severe factor V deficiency presenting as subdural haematoma in the newborn. Eur J Pediatr. 1998 Dec;157(12):1032. doi: 10.1007/s004310050993. No abstract available. PMID 9877047
- [Result] Kulkarni R, Soucie JM. Pediatric hemophilia: a review. Semin Thromb Hemost. 2011 Oct;37(7):737-44. doi: 10.1055/s-0031-1297164. Epub 2011 Dec 20. PMID 22187396
- [Result] von der Lippe C, Frich JC, Harris A, Solbraekke KN. Treatment of hemophilia: A qualitative study of mothers' perspectives. Pediatr Blood Cancer. 2017 Jan;64(1):121-127. doi: 10.1002/pbc.26167. Epub 2016 Jul 29. PMID 27472376
- [Result] KENDALL AG, LOWENSTEIN L. Alterations in blood coagulation and hemostasis during extracorporeal circulation. II. Can Med Assoc J. 1962 Oct 20;87(16):859-64. No abstract available. PMID 14031889